CLINICAL TRIAL: NCT03848299
Title: Personalized Nutrition & Citizen Science: A Healthy Diet Through Algorithms
Brief Title: Food & You: A Healthy Diet Through Algorithms
Acronym: FoodAndYou
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Principal Investigator, Marcel Salathé, Associate Professor, Ecole Polytechnique Fédérale de Lausanne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-02124
Record Dates: First submitted 2019-02-12; First posted 2019-02-20 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Food Habits
Keywords: Glycemic responses; Microbiota; Personalized nutrition; Digital cohort; Citizen Science
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: The objective is to investigate the post-meal glucose response variations between individuals in function of their individual factors such as their microbiome composition or their lifestyle.
  All participants of the main cohort will have to follow a standardized diet during the first meal of the day from the second to the seventh day of the study participation.
  All participants will follow the same diet, except the ones that are intolerant or allergic to lactose or/and gluten. In those cases, they will follow an adapted diet for their intolerance or allergies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Single Arm (Experimental): All participants will have to consume the same standardized breakfasts from the second to the seventh day, except the ones that are intolerant or allergic to lactose or/and gluten. In those cases, they will follow an adapted diet for their intolerance or allergies.
  Interventions: Other: Experimental: Single Arm

INTERVENTIONS:
Other: Experimental: Single Arm — All participants will have to consume the same standardized breakfasts from the second to the seventh day, except the ones that are intolerant or allergic to lactose or/and gluten. In those cases, they will follow an adapted diet for their intolerance or allergies.
  Day 2 and 3: 110 g white bread.
  Day 4 and 5 : 110 g white bread and 30 g butter or 55 g white bread, 50 g dark chocolate for lactose intolerant.
  Day 6 and 7: Glucose drink (50g).
  The bread will be replaced by gluten-free bread for gluten intolerant participants.
  Other Names: Standardized breakfasts consumption

SUMMARY:
Food & You is a large-scale citizen science research project in Switzerland. With this project, the researchers want to confirm that individuals respond differently to food, that is, that the blood sugar response (the level of sugar in the blood after a meal) varies among individuals, even after consumption of the same food or beverage. Secondly, the researchers want to develop an algorithm that will predict the individual blood sugar response and provide personalized diet recommendations.

DETAILED DESCRIPTION:
Food & You is one of the first large-scale citizen science research project in Switzerland. This project is building on the results of Zeevi et al. study, which demonstrated in 2015 for the first time with a cohort of 800 participants that there is a high interpersonal variability in postprandial (postmeal) glycemic responses (PPGR). In a second stage, the group developed an algorithm that predicts PPGR and gives personalized diet recommendation to better control the blood sugar level. These results have only been shown once, if they turn out to be correct, it will have a very strong impact on the field of nutrition. Other studies have since then also shown the variability in glucose response, leading to the concept of individual "glucotypes". The most important particularity of Food & You is that it will be a citizen science project. Citizen science is a method that involves volunteers in scientific research activities. It increases scientific knowledge, raises people's awareness of scientific questions, and allows scientists to share enthusiasm and expertise. Furthermore, to enable any citizen to take part, the study will be entirely coordinated digitally. It means that unlike conventional studies, no face-to-face interviews or medical appointments will be organized. All instructions will be given by a website and emails / text messages sent to the participants. The study material will be sent by post and the data will be collected via the website and the MyFoodRepo app. The participants will have to track during 14 days:

* Their dietary intake with the myFoodRepo app.
* Their physical activity and sleep with a smartphone app or an activity tracker.
* Their glucose level wearing the FreeStyle Libre Sensor.
* Collect a stool sample. The microbiome composition will be analyzed by sequencing the 16s rDNA extracted from the stool sample.
* Answer anthropometric, demographic, and health online questionnaires.

With the Food & You project, the research team will build a new algorithm that will predict PPGR with input that is readily available through such a "digital cohort" (i.e. low-burden on user, and affordable) in order to test whether this can scale to tens or hundreds of thousands of people. The results of this project may have substantial consequences in dietary guidelines, personalized diet and on health conditions related to dietary intake.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18+.
* Have a postal address in Switzerland.
* Own a smartphone, minimum version iOS 10/Android 5.
* Sufficient knowledge of French, German or English to read and understand the instructions.
* Able to provide an informed consent.

Exclusion Criteria:

* Pregnancy.
* Persons on dialysis.
* Persons with chronic immunosuppressive medication usage.
* persons with skin disease, including contact dermatitis
* Critically-ill patients.
* Breastfeeding.
* Usage of antibiotics in the three months prior to enrollment.
* Chronically active inflammatory or neoplastic disease in the three years prior to enrollment.
* Chronic gastrointestinal disorder, including Inflammatory Bowel Disease and Celiac disease.
* Active neuropsychiatric disorder.
* Myocardial infarction or cerebrovascular accident in the six months prior to enrollment.
* Pre-diagnosed type I or type II diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 50% men, 50% women
Enrollment: 1782 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Blood glucose level | Two weeks
  The participants will use the Flash Glucose Monitor FreeStyle Libre sensor and the FreeStyle Libre smartphone app from Abbott Diabetes Care to measure continuously during 14 days their glucose level.

SECONDARY OUTCOMES:
Dietary intake | Two weeks
  Food consumption information will be collected through the smartphone app myFoodRepo. The participants will track their dietary intake by taking pictures of all consumed food and beverages (including water).
Physical activity intensity | Two weeks
  The intensity of the physical activity. By default, the participants will have to log manually this features in the study website. In case a participant prefers to use an activity tracker or a smartphone app he/she owns instead of manual logging, it will also be possible.
Physical activity frequency | Two weeks
  The frequency of the physical activity. By default, the participants will have to log manually this features in the study website. In case a participant prefers to use an activity tracker or a smartphone app he/she owns instead of manual logging, it will also be possible.
Physical activity duration | Two weeks
  The duration of the physical activity. By default, the participants will have to log manually this features in the study website. In case a participant prefers to use an activity tracker or a smartphone app he/she owns instead of manual logging, it will also be possible.
The sleep duration | Two weeks
  The duration of sleep will be assessed. By default, the participants will have to log manually this features in the study website. In case a participant prefers to use an activity tracker or a smartphone app he/she owns instead of manual logging, it will also be possible.
The sleep timing | Two weeks
  The timing of sleep will be assessed. By default, the participants will have to log manually this features in the study website. In case a participant prefers to use an activity tracker or a smartphone app he/she owns instead of manual logging, it will also be possible.
Microbiome composition | Once during the two weeks
  The participants will collect a stool sample. We will transfer the samples to Microsynth, a company specialized in DNA sequencing. They will extract the DNA from the stool sample and sequence the ribosomal DNA (16S rDNA) with Next-Generation Sequencing (NGS) technology. The composition of microbial communities in the gut of each participant will be determined by bioinformatic analysis.
Optional: menstrual cycle ovulation day | Four weeks
  The ovulation day will be detected by basal temperature measurements and optionally the cervical mucus quality observations. The participants will have to log manually this features in the study website. This part is optional.
Optional: the pain related to the premenstrual syndrome (PMS) | Four weeks
  The pain will be assessed to detect PMS. The participants will have to log manually this features in the study website. This part is optional.
Optional: the quality of digestion related to the premenstrual syndrome (PMS) | Four weeks
  The quality of digestion will be assessed to detect PMS. The participants will have to log manually this features in the study website. This part is optional.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Salathé, Pr, Principal Investigator — Ecole Polytechnique Fédérale de Lausanne
Locations (1):
- Epfl Sv Ghi Upsalathe1, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh R, McDonald D, Hernandez AR, Song SJ, Bartko A, Knight R, Salathe M. Temporal nutrition analysis associates dietary regularity and quality with gut microbiome diversity: insights from the Food & You digital cohort. Nat Commun. 2025 Sep 30;16(1):8635. doi: 10.1038/s41467-025-63799-z. PMID 41028733